CLINICAL TRIAL: NCT07293156
Title: Impact of Pilates Exercises on Diabetic Erectile Dysfunction.
Acronym: PilatesDED2025
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Collaborators: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mahmoud Hamada Mohamed, Associate Professor of Physical Therapy, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pilate Exercises for DED2025
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Diabete Mellitus; Erectile Dysfunction Associated With Type 2 Diabetes Mellitus; Pilates Exercise; Pelvic Floor Muscle Exercise
Keywords: Diabete Mellitus; Erectile dysfunction; Pilates exercises; Pelvic floor exercises
MeSH Terms: conditions — Diabetes Mellitus; Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Interventional
Who Masked: Participant
Masking Description: Single (Participant) This is a parallel group randomized controlled trial with two arms receiving different interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): study group
  Interventions: Other: Pilate Exercises; Other: Pelvic floor muscles exercises
- Active comparator (Active Comparator): control
  Interventions: Other: Pelvic floor muscles exercises

INTERVENTIONS:
Other: Pilate Exercises — Pilates protocol that will be used in the present study consisted of 11 different Pilates postures: Pilates Breathing, Spine Stretch, Swan, Shoulder Bridge, Hundreds, Double Leg Stretch, Footwork, Roll up, Single Leg Stretch, Leg Pull Back, Kick front and back. It will be performed thrice a week, with each session lasting 60 minutes, for 12 weeks, totaling 36 sessions. The progression of the exercises will be based on increasing the number of repetitions of the exercise, and variations in posture from beginner to intermediate and advanced, for each exercise. The movements will be repeated six to eight times each.
  Arms: Experimental
Other: Pelvic floor muscles exercises — The pelvic floor exercises will be taught by a skilled physiotherapist who instructed the men to tighten their pelvic floor muscles as strongly as possible (as if to prevent flatus from escaping), to gain muscle hypertrophy. During pelvic floor muscle training attention was placed on the ability to retract the penis and lift the scrotum, to make sure the bulbocavernosus and ischiocavernosus muscles were working strongly. Emphasis was placed on gaining a few maximum contractions (three when lying, three sitting, and three standing) twice daily rather than prolonged repetitions. Some submaximal pelvic floor work will be advised while walking, to increase muscle endurance. Men will be also taught to tighten their pelvic floor muscles strongly after voiding urine whilst still poised over the toilet, as a way of working the bulbocavernosus muscle to eliminate the urine from the bulbar urethra.
  Frequency of treatment: Treatment will be given 3 times / week for 12 weeks total of 36 session

SUMMARY:
Erectile dysfunction (ED) has a prevalence of 52.5% in diabetic male patients, as described in a meta-analysis of 145 studies, including 88,577 men with type 1 and type 2 diabetes.

In men, ED can cause sexual dissatisfaction and distress, unsatisfactory relationships, and marital tension

DETAILED DESCRIPTION:
Pilates emerged as a method of rehabilitation during World War I, when Joseph Hubertus Pilates applied his knowledge to rehabilitate injured men. The popularity of the method grew most in the 1980. More recently, Pilates has been used resulting in improved fitness (flexibility, strength and balance) and body consciousness. The method features ground-based exercises created by Joseph Pilates.

Because most Pilates exercises are performed in conjunction with the recruitment of PF muscle fibres, many Pilates instructors believe that the method can produce a significant increase in the force or contractility of the muscles. Furthermore, if Pilates promotes an improvement in the functioning of the pelvic floor muscles (PFM), it may be an alternative for the treatment and prevention of pelvic floor dysfunction.

Up till now, no published trials about impact of Pilate exercises on diabetic erectile dysfunction.

A total of 60 patients (n=30 per group), diagnosed with diabetic erectile dysfunction in the past 6 months. Participants will be recruited from Benha University hospital and local andrology and urology clinics in benha and giza . Participants will be screened for eligibility prior to being enrolled in the study participating in the study assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 40-60 years.
2. Diagnosed diabetes mellitus (type 2) ≥ 1 year.
3. Clinical diagnosis of erectile dysfunction for ≥ 6 months, confirmed by IIEF5 score.
4. Stable antidiabetic medications for ≥ 3 months prior to randomization.
5. HbA1c between 6.5% and 10.0%.
6. Sexually active or attempting sexual activity at least occasionally (at least once monthly) and willing to attempt intercourse during study.
7. Able and willing to participate in the exercise program (physically capable and available for scheduled sessions) and provide written informed consent.

Exclusion Criteria:

1. Severe cardiovascular disease within past 6 months (e.g., recent myocardial infarction, unstable angina, decompensated heart failure, uncontrolled arrhythmia) that contraindicates exercise.
2. Uncontrolled hypertension (e.g., systolic ≥ 180 mmHg or diastolic ≥ 110 mmHg) despite treatment.
3. Severe peripheral vascular disease or other conditions preventing safe exercise (severe claudication, severe orthopedic limitations).
4. History of pelvic surgery or pelvic radiation within the last 12 months that could acutely affect erectile function.
5. Primary neurogenic causes of ED unrelated to diabetes (spinal cord injury, multiple sclerosis).
6. Major psychiatric illness or severe cognitive impairment interfering with consent/compliance .
7. Current substance abuse or heavy alcohol use that could affect sexual function or compliance.
8. Severe hypogonadism requiring imminent testosterone therapy (total testosterone < 8 nmol/L with symptoms).
9. Active genitourinary infection or untreated severe sexual dysfunction disorders other than ED.
10. Use of medications known to cause ED that cannot be discontinued or stabilized.
11. Current participation in structured pelvic floor or sexual-function exercise program similar to the intervention.
12. Recent (within 4 weeks) or planned changes in PDE5i therapy.
13. Any medical condition making participation unsafe or likely to confound outcomes per investigator judgment.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Males with diabetic erectile dysfunction
Enrollment: 60 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
penile perfusion | Base line and after 12 weeks
  Colour-coded duplex sonography (5-10 MHz probes) will be used for the evaluation of penile perfusion. Half ml of a vasoactive agent (trimix solution) will be injected into the corpus cavernosum. The systolic and diastolic velocities (cm/s) will be performed at 10 and 30 min for both cavernous artery. Re-dosing with 0.5 ml of trimax solution will be performed for patients who did not achieve adequate hardness. The highest values obtained will be recorded. The following Doppler indices of the right and left cavernous arteries: peak systolic velocity (PSV), end-diastolic velocity (EDV) and resistance index (RI) will be recorded.

SECONDARY OUTCOMES:
International Index of Erectile Function-5 (IIEF-5) scale. | Baseline and after 12 weeks
  The IIEF-5 scale is used to assess patients with erectile dysfunction to determine the extent of the erectile function in patients. The full-scale 15-item version has five domains: erectile function, orgasmic function, sexual desire, intercourse satisfaction and overall sexual satisfaction.
  The shortened 5-item version is on a scale of 5 to 25:
  22-25: No erectile dysfunction 17-21: Mild erectile dysfunction 12-16: Mild to moderate erectile dysfunction 8-11: Moderate erectile dysfunction 5-7: Severe erectile dysfunction

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Outpatient clinic, faculty of Physical Therapy, Benha university, Banhā, Benha
  - Outpatient clinic, faculty of Physical Therapy, Ahram Canadian university, Giza, Giza Governorate

IPD SHARING:
Plan to Share IPD: Undecided